CLINICAL TRIAL: NCT04061135
Title: Neurophysiological, Behavioral, and Cognitive Networks in Movement Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, J. Nicole Bentley, Principle Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300003605; UAB (Other: UAB)
Record Dates: First submitted 2019-07-16; First posted 2019-08-19 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Movement Disorders
Keywords: Parkinson's disease
MeSH Terms: conditions — Movement Disorders; Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Parkinson's Disease Patients receiving DBS electrodes
  Interventions: Procedure: Response Inhibition and Deep Brain Stimulation in Parkinson's disease
- Control (No Intervention): Control subjects will be non-Parkinson's Disease patients with essential tremor

INTERVENTIONS:
Procedure: Response Inhibition and Deep Brain Stimulation in Parkinson's disease — After creation of the burr hole and prior to DBS electrode placement, 1-2 subdural strip electrodes will be placed anteriorly or posteriorly from the cranial opening. These electrodes are routinely placed using this technique for seizure mapping, with arrays of electrodes (up to 6) being placed around the perimeter of the opening.14 Subdural strips vary in length and contact size (e.g., the 6-contact Ad-Tech strip), and are currently placed predominantly for studies of sensorimotor function,13 including at our institution (IRB-140327003). Placement over prefrontal areas is performed at other institutions.11-13 The DBS surgery will then proceed according to routine practice, and following lead placement in the optimal desired location, the research task paradigm will begin.
  Arms: Treatment

SUMMARY:
The purpose of this study is to investigate the brain activity associated with motor and non-motor symptoms of movement disorders, including Parkinson's disease (PD) and essential tremor. These movement disorders commonly have significant non-motor features, such as depression, cognitive and memory impairment, decreased attention, speech and language disturbances, and slower processing speeds. The investigators are interested in the brain activity associated with these motor and non-motor symptoms, and propose to investigate changes in brain activity while the investigators perform recordings of the surface and deep structures of the brain, in addition to the typical recordings the investigators perform, during routine deep brain stimulation (DBS) surgery.

DETAILED DESCRIPTION:
Movement disorders are a prominent cause of disability worldwide. In the United States, it is estimated that more than 4 million people suffer from Parkinson's disease (PD), essential tremor (ET), and dystonia, making them some of the most prevalent of neurologic disorders. Of these, PD is the most common, and is primarily characterized by tremor, rigidity, and bradykinesia. However, though primarily characterized by motor symptoms, many patients also have prominent non-motor features, including depression and cognitive impairment, with deficiencies in processing speed, memory, attention, and learning. Some of the most debilitating cognitive deficiencies include deficits in goal-directed response selection and response inhibition, language, and/or speech difficulties, all of which substantially contribute to reduced quality of life.

Unfortunately, these features of movement disorders are less well-studied and lack effective treatment options, necessitating that new treatments be investigated. Deep brain stimulation (DBS), while a highly effective treatment for the cardinal features of PD, is essentially ineffective for, and can even worsen other cognitive domains, and there are few studies currently investigating how different parameters of DBS may improve these symptoms. In addition, speech abnormalities are common with Parkinson's disease and DBS can sometimes worsen speech problems. These impairments consists primarily of hypophonia, but cognitive deficits can result in actual language disturbance. It is often difficult to know whether the speech problems are related to language processing or articulation (related to the movement disorder). In an effort to begin addressing these questions, we propose to study motor and non-motor symptoms in patients with movement disorders, and to correlate movement and cognition with underlying neural electrophysiology.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for DBS surgery based on multi-disciplinary consensus review
* Have a diagnosis of Parkinson's disease or Essential Tremor
* A minimum of 18 years of age
* Willingness to participate in the paradigms described in the protocol

Exclusion Criteria:

* Inability to provide full and informed consent
* Are not surgical candidates due to co-morbid conditions or pregnancy
* Have not undergone an adequate trial of conservative medical management
* Have a clinical presentation for which DBS surgery is not indicated
* Are not able to participate in study-related activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy via Simon Task (% correct) | Baseline
  In the Simon task, participants are instructed to respond with a right or left button press (Right = Red, Left = Blue) according to how a word is printed on a screen ("RED" or "BLUE"), regardless of the color in which the word is printed.
  This is a measurement of accuracy (% correct, ranging from 0-100, with higher scores indicating better performance)
Response times via Simon Task (sec) | Baseline
  In the Simon task, participants are instructed to respond with a right or left button press according to the word "RIGHT" or "LEFT" that appears on a screen, regardless of where on the screen it actually appears.
  This is a measurement response times (continuous measure, from 0-4000 milliseconds) between correct and incorrect responses.
Simon Effect on Response times (sec) | Baseline
  Participants will perform the Simon task as described, and the Simon effect will be calculated as the difference in response times between congruent and incongruent trials
Simon Effect on Accuracy (% correct) | Baseline
  Participants will perform the Simon task as described, and the Simon effect will be calculated as the difference in accuracy between congruent and incongruent trials
UPDRS 3 motor score (0-108) | Baseline
  Participants will undergo motor evaluation using the validated United Parkinson's disease Rating Scale (UPDRS) part 3
Dementia Rating Scale Score (0-144 points) | Baseline
  Participants will undergo neuropsychological testing as part of routine care, including the Dementia Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Bentley, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No